CLINICAL TRIAL: NCT03908879
Title: Prospective Diagnostic Accuracy Study Comparing Sensitivity and Specificity of Methods Used to Confirm Correct Placement of an Intraosseous (IO) Catheter
Brief Title: Intraosseous Catheter Confirmation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Yonatan Greenstein, MD, Associate Professor of Medicine, Division of Pulmonary & Critical Care Medicine, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro2019000600
Record Dates: First submitted 2019-04-04; First posted 2019-04-09 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Critical Illness
Keywords: Intraosseous catheter; Intraosseous access; Resuscitation; Diagnostic accuracy
MeSH Terms: conditions — Critical Illness | interventions — Jupiter

STUDY DESIGN:
Intervention Model Description: All study participants will undergo all confirmation tests
Masking Description: There is only one arm because all participants will be undergoing the same protocol. To evaluate inter-operator variability for methods 2 and 3, co-investigators will be reviewing saved images recorded by the physicians who placed the intraosseous (IO) catheter. Saved images include the color flow Doppler image for method 2 and the pressure waveform for method 3. Two co-investigators will review saved images from method 2, blinded and independently. Two other co-investigators will review saved images from method 3, blinded and independently. If the results of the two co-investigators for method 2 or method 3 is discordant then a third blinded reviewer will review the saved image for the method with discordant results.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intraosseous (IO) catheter placement confirmation methods (Experimental): All patients will undergo all three confirmation methods/procedures. Method 1 is a triage test and an index test. Method 2 is an index test. Method 3 is a reference standard. None of the procedures being performed in this study are regulated by the United States Food and Drug Administration.
  Interventions: Procedure: Standard intraosseous (IO) catheter confirmation procedure; Procedure: Color flow Doppler intraosseous (IO) catheter confirmation procedure; Procedure: Pressure transduction intraosseous (IO) catheter confirmation procedure

INTERVENTIONS:
Procedure: Standard intraosseous (IO) catheter confirmation procedure — The physician will evaluate the ability or inability of the intraosseous (IO) catheter to stand upright unassisted, the ability or inability to aspirate blood or bone marrow from the IO catheter, and whether or not there is visible or palpable extravasation of infusate from the IO catheter insertion site or surrounding subcutaneous tissue during IO catheter use.
  Other Names: Method 1
Procedure: Color flow Doppler intraosseous (IO) catheter confirmation procedure — The high frequency probe of a portable ultrasound with color flow Doppler is placed adjacent to the intraosseous (IO) catheter, visualizing the IO space in long or short axis. Color flow Doppler signal will be turned on during IO use and the physician will determine if the Doppler signal is in the intraosseous space or the extraosseous space. Saved data of the ultrasound image will be reviewed independently by at least two blinded reviewers. If the conclusions from the blinded reviewers are discordant then a third blinded reviewer will evaluate the saved data.
  Other Names: Method 2
Procedure: Pressure transduction intraosseous (IO) catheter confirmation procedure — The intraosseous (IO) catheter will be attached to a pressure transducer to demonstrate a waveform on the telemetry monitor. Physicians will evaluate for the presence of a pulsatile waveform with objective measurements of a systolic pressure, diastolic pressure and mean pressure. Saved data of the waveform image will be reviewed independently by at least two blinded reviewers. If the conclusions from the blinded reviewers are discordant then a third blinded reviewer will evaluate the saved data.
  Other Names: Method 3

SUMMARY:
This is a prospective diagnostic accuracy study investigating the sensitivity and specificity of methods used to confirm correct placement of an intraosseous (IO) catheter. Intraosseous catheters allow medical providers to rapidly administer fluids and medications to critically ill patients when intravenous (IV) access is not present or difficult to achieve. It is standard of care to confirm the correct placement of an IO catheter prior to using it to administer medications or fluids. Three IO placement confirmatory tests will be performed on all research subjects using a standardized protocol. There will be two index tests (the method utilized by most of the medical community evaluating the stability of the catheter, ability to aspirate blood or bone marrow and ability to administer fluids without visible or palpable extravasation as well as the method of demonstrating color flow Doppler only within the intraosseous space during bedside ultrasound exam) and one reference test (ability to visualized a pulsatile waveform when the IO catheter is attached to a pressure transducer). Primary outcome measures of the study will be the determination of correct or incorrect IO catheter placement from the confirmation methods. This data will be used to investigate the primary endpoints of sensitivity and specificity of the confirmation tests as well as inter-operator variability interpreting the raw data from the confirmation methods. Secondary outcomes include complications from the IO catheter. The goal of this study is to see if a more sensitive and specific method of IO catheter confirmation can reliably be performed by different physicians and reduce the amount of complications associated with the catheters. Additional subgroup analyses will be performed in regards to the research subjects BMI and the anatomic site selected for IO catheter use (proximal tibia or humeral head).

ELIGIBILITY:
Inclusion Criteria:

* Patients greater than 18 years of age
* Full code
* Require placement of an intraosseous catheter for emergent resuscitation due to lack of reliable intravenous access
* Capable of undergoing all three intraosseous placement confirmatory methods

Exclusion Criteria:

* Age less than 18 years old
* Pregnant patients
* Prisoner/incarcerated
* Patients unable to undergo all three intraosseous placement confirmatory methods

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-07-23 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Categorical determination of correct IO catheter placement by physicians placing the catheter | Within 24 hours of intraosseous (IO) catheter insertion
  Categorical determination (yes/no) regarding correct IO catheter placement in the intraosseous space of all three confirmatory methods from the physicians placing the IO catheter
Categorical determination of correct IO catheter placement by blinded reviewers | Within 1 week of ultrasound images and pressure transduction images being created by the physician placing the IO catheter
  Categorical determination (yes/no) regarding correct IO catheter placement in the intraosseous space for method 2 and method 3 by the blinded reviewers

SECONDARY OUTCOMES:
IO catheter pressure | Within 24 hours of intraosseous (IO) catheter insertion
  Pressures measured from transducing the IO catheter: systolic pressure, diastolic pressure, mean pressure
Systemic blood pressure | Within 24 hours of intraosseous (IO) catheter insertion
  Pressures measured from a noninvasive blood pressure cuff or an arterial line: systolic pressure diastolic pressure mean pressure
Number of attempts to place IO catheter | Within 24 hours of intraosseous (IO) catheter insertion
  Number of attempts made to place an IO catheter
Complications related to IO catheter | Within 28 days of IO catheter insertion
  Complications associated with the IO catheter after insertion

CONTACTS AND LOCATIONS:
Overall Officials: Yonatan Greenstein, MD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- University Hospital, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stone MB, Teismann NA, Wang R. Ultrasonographic confirmation of intraosseous needle placement in an adult unembalmed cadaver model. Ann Emerg Med. 2007 Apr;49(4):515-9. doi: 10.1016/j.annemergmed.2006.11.009. Epub 2007 Jan 12. PMID 17222940
- [Background] Tsung JW, Blaivas M, Stone MB. Feasibility of point-of-care colour Doppler ultrasound confirmation of intraosseous needle placement during resuscitation. Resuscitation. 2009 Jun;80(6):665-8. doi: 10.1016/j.resuscitation.2009.03.009. Epub 2009 Apr 22. PMID 19395142
- [Background] Frascone RJ, Salzman JG, Ernest EV, Burnett AM. Use of an intraosseous device for invasive pressure monitoring in the ED. Am J Emerg Med. 2014 Jun;32(6):692.e3-4. doi: 10.1016/j.ajem.2013.12.029. Epub 2013 Dec 18. PMID 24440591
- [Background] Salzman JG, Loken NM, Wewerka SS, Burnett AM, Zagar AE, Griffith KR, Bliss PL, Peterson BK, Ward CJ, Frascone RJ. Intraosseous Pressure Monitoring in Healthy Volunteers. Prehosp Emerg Care. 2017 Sep-Oct;21(5):567-574. doi: 10.1080/10903127.2017.1302529. Epub 2017 Apr 18. PMID 28418753
- [Derived] Greenstein YY, Ferrara S, Jomi J, Soetanto V, Zuckerman O, Sena A, Ostrovsky I, Alerhand S. A Prospective Comparison of Standard Technique, Doppler Ultrasonography, and Pressure Waveform Analysis for Confirming Intraosseous Catheter Placement. J Intensive Care Med. 2024 Mar;39(3):222-229. doi: 10.1177/08850666231199086. Epub 2023 Aug 30. PMID 37647305